CLINICAL TRIAL: NCT03364777
Title: Analysis of Correlations Between Preoperative Emotional State and Postoperative Clinical Effect in Patients Undergoing Lumbar Surgery
Brief Title: The Correlations Between Clinical Effect and Emotional State
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Chenjun, spinal surgery, Peking University People's Hospital
Other Study IDs: Emotionalstate
Record Dates: First submitted 2017-11-26; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Emotional Disorder
Keywords: lumbar surgery, emotional state
MeSH Terms: interventions — Mental Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lumbar surgery patients: patients undergoing lumbar surgery with or without anxiety or depression emotional state
  Interventions: Other: emotional state

INTERVENTIONS:
Other: emotional state — anxiety or depression state evaluated by emotional scale

SUMMARY:
To analyze the correlations between preoperative emotional state and postoperative clinical effect among patients undergoing lumbar surgery

DETAILED DESCRIPTION:
Preoperative emotional state and postoperative clinical effect of patients undergoing lumbar surgery will be evaluated and compared. Then the relations of anxiety and depression on quality of life will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. patients with relevant symptoms of lumbar degenerative diseases;
2. patients with bad emotional state,such as anxiety or depression.

Exclusion Criteria:

1. spinal tumor;
2. spinal trauma;
3. congenital spinal disease;
4. patients diagnosed psychosis;
5. patients with incomplete clinical informations.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing lumbar surgery for lumbar degenerative diseases with or without emotional state of anxiety and depression evaluated by emotional scales.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
changes of patient's quality of life | Baseline and two weeks postoperative
  difference of scores of clinical effect scales

SECONDARY OUTCOMES:
changes of patients's emotional state | Baseline and two weeks postoperative
  difference of scores of emotional state scales

CONTACTS AND LOCATIONS:
Overall Officials: Haiying Liu, doctor, Study Director — spinal surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Floyd H, Sanoufa M, Robinson JS. Anxiety's Impact on Length of Stay Following Lumbar Spinal Surgery. Perm J. 2015 Fall;19(4):58-60. doi: 10.7812/TPP/15-022. PMID 26517435
- [Background] Falavigna A, Righesso O, Teles AR, Baseggio N, Velho MC, Ruschel LG, Abruzzi F, Silva PG. Depression Subscale of the Hospital Anxiety and Depression Scale applied preoperatively in spinal surgery. Arq Neuropsiquiatr. 2012 May;70(5):352-6. doi: 10.1590/s0004-282x2012000500009. PMID 22618787
- [Background] D'Angelo C, Mirijello A, Ferrulli A, Leggio L, Berardi A, Icolaro N, Miceli A, D'Angelo V, Gasbarrini G, Addolorato G. Role of trait anxiety in persistent radicular pain after surgery for lumbar disc herniation: a 1-year longitudinal study. Neurosurgery. 2010 Aug;67(2):265-71. doi: 10.1227/01.NEU.0000371971.51755.1C. PMID 20644411